CLINICAL TRIAL: NCT00511446
Title: Phase II Trial of Docetaxel, Oxaliplatin and Capecitabine (TEX) in Advanced or Metastatic Gastric Cancer
Brief Title: Trial of Docetaxel, Oxaliplatin and Capecitabine (TEX) in Advanced or Metastatic Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Hans-Joachim Schmoll, MD, MD, Martin-Luther-Universität Halle-Wittenberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIO STO-0601
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Stomach Neoplasms
Keywords: Stomach neoplasms; docetaxel; oxaliplatin; capecitabine
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): docetaxel, oxaliplatin, capecitabine
  Interventions: Drug: docetaxel, oxaliplatin, capecitabine

INTERVENTIONS:
Drug: docetaxel, oxaliplatin, capecitabine — Docetaxel: 35 mg/m2, IV day 1, 8 of each 21 day cycle; Oxaliplatin: 70 mg/m2, IV day 1, 8 of each 21 day cycle; Capecitabine: 2x800 mg/m2 PO IV day 1 evening till morning of day 15 of each 21 day cycle.
  Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: xeloda; taxotere; eloxatin

SUMMARY:
Combination regimens of 3 active drugs have shown promising activity in treatment of metastatic gastric cancer. Docetaxel combined with cisplatin and 5-fluorouracil (FU) yielded superior overall survival and response rates when compared to standard cisplatin and 5-FU. However, a toxicity profile showed the need for development of less toxic modifications. In a prior phase I trial, the maximum tolerated dose was defined. In this phase II trial, a first evaluation of activity will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Histologically proven irresectable, metastatic or recurrent adenocarcinoma of the stomach or the gastroesophageal junction, i.e., Tx-4 M1 or T4 M0
* Irresectable (as judged by an experienced surgeon):

  1. T4 infiltrating of several organs
  2. T4 infiltrating one organ, but irresectable
  3. T4 infiltrating one organ, respectable, but inoperable patient
* The nodal status is neglected
* Measurable disease according to RECIST
* ECOG Performance Status ≤ 2
* Male or female patients aged ≥ 18 years
* Life expectancy ≥ 3 months
* Adequate bone marrow, hepatic and renal function:

  1. Haemoglobin > 9.0 g/dL (transfusions allowed to achieve or maintain levels)
  2. Absolute neutrophil count > 1.5 x 10^9/L
  3. Platelet count > 100 x 10^9/L
  4. ALAT, ASAT < 3.5 x ULN
  5. Alkaline phosphatase < 6 x ULN
  6. Total bilirubin < 1.0 x ULN
  7. Creatinine clearance > 50 mL/min (calculated according to Cockroft and Gault)
* Prior surgery must be more than 28 days ago
* Positive nodes as diagnosed on endorectal ultrasound and/or MRI (tumour is staged by preferably a high resolution MRI; if MRI is not available, locoregional staging must be performed by computed tomography plus endorectal ultrasound)
* Tumor staging must be done within 28 days from the start of the treatment
* Negative pregnancy test in women with childbearing of potential (within 7 days prior to the start of the chemotherapy)

  * Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential

Exclusion Criteria:

* Prior cytotoxic chemotherapy or radiotherapy (a neoadjuvant or adjuvant chemotherapy must be completed and without progression for at least 6 months)
* Previous (within the last 5 years) or concurrent malignancies, with the exception of adequately treated in situ carcinoma of the cervix or basal cell carcinoma of the skin
* Peripheral neuropathy ≥ grade 2 (according to NCI CTCAE v 3.0)
* Patient must not have been treated with any investigational drug, agent nor procedure, (i.e., did not participate in another trial within 30 days) before entry in this trial
* Known allergy or any other adverse reaction to any of the study drugs or to any related compound
* Requirement for concurrent use of the antiviral agent sorivudine (antiviral) or chemically related analogues, such as brivudine
* Clinically significant concomitant diseases, such as:

  1. Active infection necessitating systemic antibiotics
  2. Interstitial lung diseases
  3. Chronic diarrhea, inflammatory bowel disease
  4. Neurological or psychiatric disease, dementia, epilepsy or untreated brain metastases
* Cardiac disease (e.g., congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmia not well controlled with medication) or myocardial infarction or resuscitation within the last 6 months
* Pregnant or lactating women are excluded
* Presence of adequate contraception in fertile patients (methods of adequate contraception are: intra-uterine device, hormonal contraception, vasectomy, tubal ligation or abstinence)
* Alcohol or drug abuse
* Ability to swallow tablets
* Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-08; Primary Completion 2010-05 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival rate | at 6 months

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety/toxicity | 2 years
Median time to progression | 2 years
Response rate | 2 years
Rate of resections with curative intent | 2 years
Time to treatment failure | 2 years
Duration of response | 2 years
Median overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Joachim Schmoll, Prof. Dr., Principal Investigator — Martin-Luther-University Halle-Wittenberg, Medical Faculty
Locations (10):
- Germany (10):
  - Charite - Universitatsmedizin Berlin, Berlin
  - Medizinische Universitätsklinik - Knappschaftskrankenhaus, Bochum
  - Städtische Kliniken Esslingen, Esslingen am Neckar
  - MVZ Osthessen, Fulda
  - Martin-Luther-University Halle-Wittenberg, Halle
  - Städt. Klinikum St. Georg, Leipzig
  - OSP Lörrach-Rheinfelden, Loerrach
  - Universitätsklinikum Mainz, Mainz
  - Universitätsklinikum Mannheim, Mannheim
  - Universitätsklinik Ulm, Ulm

REFERENCES:
- See also: Arbeitsgemeinschaft Internistische Onkologie — http://www.aio-portal.de